CLINICAL TRIAL: NCT03008057
Title: The Assessment of the Effect of Vitamin D Supplementation on the Serum of AGES and Endothelialy Factors and Gene Expression of Glyoxalase Enzyme and YKL-40 Factor in PBMC Cells in the Patients With Type 2 Diabetes .
Brief Title: The Assessment of the Effect of Vitamin D Supplementation on Inflammatory and Endothelial Factors in the Patients With Type 2 Diabetes .
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 32615
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes
Keywords: vitamin D; YKL40; PAI-1; RAGE; AGEs; glyoxalase enzyme; TNF-alpha; IL-6; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D supplementation (Active Comparator): patients with type 2 diabetes receive 1 tablet (4000 IU ) vitamin D supplementation, one time a day, for 3 months.
  Interventions: Dietary Supplement: vitamin D
- vitamin D placebo (Placebo Comparator): patients with type 2 diabetes receive one tablet of vitamin D placebo for 3 months
  Interventions: Dietary Supplement: vitamin D placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — vitamin D supplement, 4000 IU tablet daily , one time a day, for 3 months
  Arms: vitamin D supplementation
Dietary Supplement: vitamin D placebo — vitamin D placebo tablet (Containing starch powder), one time a day, for 3 months
  Arms: vitamin D placebo

SUMMARY:
The aim of this study is to determine the effects of vitamin D or placebo for 3 months on the gene expression of glyoxalase enzyme, RAGE, and YKL40 in the peripheral blood mononuclear cell (PBMC) and serum levels of YKL40,AGEs, TNF-α, PAI-1, IL-6, and HbA1c of diabetes type 2 patients.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of vitamin D or placebo for 3 months on the gene expression of plasma human cartilage glycoprotein 39(YKL40), receptor for advanced glycation end products (RAGE) and glyoxalase enzyme in the peripheral blood mononuclear cell (PBMC) and serum levels of YKL40 ,plasminogen activator inhibitor-1 (PAI-1), TNF-α, advanced glycation end products (AGEs ), IL-6, and HbA1c of diabetes type 2 patients.

In this randomized, double-blind clinical trial, placebo-controlled study, 84 women and men with type 2 diabetes are enrolled from the Iranian Center of diabetes. At the start of study, all participants will sign informed consent and complete a general information form. 24-hour food record for 3 days will be taken from the patients at the beginning and the end of the study. Selected samples by using stratified randomization method based on sex, gender and body mass index (BMI) are classified into 2 groups: 1) receiving vitamin D supplement 2) receiving vitamin D placebo bo.

The vitamin D supplement group will receive 4000 IU (100 microgram) daily for 3 months. The vitamin D placebo group will also receive placebo containing starch both similar in terms of color, shape and size. participants are advised to maintain their diet, level of physical activity and medication dose during the study. Blood samples will be collected after anthropometric parameter measuring then target biochemical parameters, gene expression and serum levels and physical activity will be measured before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

- diabetic type 2 patients 35-65 years old, body mass index in the range 18.5- 30 ,literate, willingness to participation,avoidance of dietary supplements, vitamins and herbal products at least 3 months before and throughout the intervention -

Exclusion Criteria:

* people who have used vitamin D supplements in last 3 months, having chronic renal disease , GI disease, Hepatobilliary diseases, hematological disorders, hypo- or hyperthyroidism, treatment with orlistat or sibutramine for weight loss, pregnancy and lactation, treatment with insulin or Thiazolidinediones, Smokers,sever change in regular diet and life style,change in type and dosage of regular medication (s)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
serum HbA1c | Change frome baseline at 3 months
serum fasting insulin | Change frome baseline at 3 months
serum Fasting blood suger, | Change frome baseline at 3 months

SECONDARY OUTCOMES:
serum AGES | Change frome baseline at 3 months
serum IL6 | Change frome baseline at 3 months
serum TNF-alpha | Change frome baseline at 3 months
serum PAI-1 | Change frome baseline at 3 months
RAGE gene expression | Change frome baseline at 3 months
YKL40 gene expression | Change frome baseline at 3 months
glyoxalase enzyme gene expression | Change frome baseline at 3 months
serum IL-17 | Change frome baseline at 3 months
Serum IL-4 | Change frome baseline at 3 months
serum Transforming growth factor beta | Change frome baseline at 3 months
serum YKL40 | Change frome baseline at 3 months

REFERENCES:
- [Derived] Omidian M, Djalali M, Javanbakht MH, Eshraghian MR, Abshirini M, Omidian P, Alvandi E, Mahmoudi M. Effects of vitamin D supplementation on advanced glycation end products signaling pathway in T2DM patients: a randomized, placebo-controlled, double blind clinical trial. Diabetol Metab Syndr. 2019 Oct 26;11:86. doi: 10.1186/s13098-019-0479-x. eCollection 2019. PMID 31673295
- [Derived] Omidian M, Mahmoudi M, Abshirini M, Eshraghian MR, Javanbakht MH, Zarei M, Hasani H, Djalali M. Effects of vitamin D supplementation on depressive symptoms in type 2 diabetes mellitus patients: Randomized placebo-controlled double-blind clinical trial. Diabetes Metab Syndr. 2019 Jul-Aug;13(4):2375-2380. doi: 10.1016/j.dsx.2019.06.011. Epub 2019 Jun 11. PMID 31405646